CLINICAL TRIAL: NCT05347225
Title: A Phase 1 Clinical Study to Investigate the Safety, Pharmacokinetics and Efficacy of MK-1026 in China Participants With Relapsed or Refractory Hematologic Malignancies
Brief Title: A Study of Nemtabrutinib (MK-1026) in China Participants With Relapsed or Refractory Hematologic Malignancies (MK-1026-005)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1026-005; MK-1026-005 (Other: MSD)
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — ARQ531

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Nemtabrutinib (Experimental): Participants receive nemtabrutinib at specified dose orally once daily (QD) until progressive disease (PD) or discontinuation.
  Interventions: Drug: Nemtabrutinib

INTERVENTIONS:
Drug: Nemtabrutinib — Nemtabrutinib tablets will be administered orally QD.
  Other Names: MK-1026; ARQ 531

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics (PK) and preliminary efficacy of oral nemtabrutinib in Chinese participants at least 18 years of age who have Relapsed/Refractory hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory participants with a diagnosis of B-cell Non-Hodgkin's Lymphoma (NHL), Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Leukemia (SLL) or Waldenström's Macroglobulinemia (WM) who have received no more than 4 prior standard systemic therapies. Participants must have failed or are intolerant to standard therapies and cannot be a candidate for standard salvage regimens and those with low grade lymphoma must be progressing and requiring treatment
* Must have received prior systemic treatment before joining this study
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* HBV/HCV viral load undetectable or no history of HBV/HCV
* Has adequate organ function
* Male participants agree to be abstinent from heterosexual intercourse or agree to use contraception during the intervention period and for at least 30 days after the last dose of the study intervention
* Female participant is not a Women of Child Bearing Potential (WOCBP) or is a WOCBP using contraception during the intervention period and for at least 30 days after the last dose of the study intervention

Exclusion Criteria:

* Has a history of prior cancer within <3 years, except for adequately treated basal cell or squamous cell carcinoma of the skin, cervical cancer in situ, or other in situ carcinomas
* Has active primary tumor involvement of central nervous system (CNS) disease
* Has an active infection requiring systemic therapy
* Has a known history of Human Immunodeficiency Virus (HIV) infection
* Has an uncontrolled illness including but not limited to ongoing symptomatic congestive heart failure (New York Heart Association Class III or IV heart failure), unstable angina pectoris, cardiac arrhythmia, and psychiatric illness
* Had immunotherapy, radioimmunotherapy, biological therapy, chemotherapy, or treatment with an investigational product ≤4 weeks prior to treatment initiation
* Has any clinically significant gastrointestinal abnormalities that might alter absorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-06-09 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who Experience Adverse Events (AEs) | Up to ~ 35 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of Participants Discontinuing Study Treatment due to AEs | Up to ~ 35 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Maximum Concentration (Cmax) of Nemtabrutinib | Day 1 of Cycles 1 and 2: Pre-dose,1, 2, 4, 6, 8, and 24 hours post-dose; Day 1 of Cycle 3: pre-dose and 2 hours post-dose (up to ~57 days). Each cycle is 28 days
  Cmax is the maximum concentration of nemtabrutinib observed in plasma. Blood samples collected at designated timepoints will be used to determine Cmax.
Minimum Concentration (Cmin) of Nemtabrutinib | Day 1 of Cycles 1 and 2: Pre-dose,1, 2, 4, 6, 8, and 24 hours post-dose; Day 1 of Cycle 3: pre-dose and 2 hours post-dose (up to ~57 days). Each cycle is 28 days
  Cmin is the minimum concentration of nemtabrutinib observed in plasma. Blood samples collected at designated timepoints will be used to determine Cmin.
Area Under the Plasma Concentration-Time Curve from 0 to 24 Hours (AUC0-24) of Nemtabrutinib | Day 1 of Cycles 1 and 2: Pre-dose,1, 2, 4, 6, 8, and 24 hours post-dose; Day 1 of Cycle 3: pre-dose and 2 hours post-dose (up to ~57 days). Each cycle is 28 days
  AUC0-24 is the area under the curve of plasma concentration of nemtabrutinib from time 0 to 24 hours. Blood samples collected at designated timepoints will be used to determine AUC0-24.
Time to Maximum Concentration (Tmax) of Nemtabrutinib | Day 1 of Cycles 1 and 2: Pre-dose,1, 2, 4, 6, 8, and 24 hours post-dose; Day 1 of Cycle 3: pre-dose and 2 hours post-dose (up to ~57 days). Each cycle is 28 days
  Tmax is the time to reach maximum concentration of nemtabrutinib. Blood samples collected at designated timepoints will be used to determine Tmax.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per International Workshop on Chronic Lymphocytic Leukemia (iwCLL) Criteria 2018 as Assessed by the Investigator | Up to ~ 35 months
  ORR per iwCLL criteria 2018 is defined as the percentage of participants achieving a complete response (CR), complete response with incomplete bone marrow (BM) recovery (CRi), nodular partial response (nPR) or partial response (PR). CR is defined as meeting the following criteria: no lymph nodes ≥1.5 cm, spleen size <13 cm, liver normal; no constitutional symptoms, normal lymphocyte count, platelets ≥100 x 10^9/L; hemoglobin ≥11 g/dL; and normocellular marrow (no CLL cells or B lymphoid nodules). CRi is defined as meeting CR criteria but with incomplete bone marrow recovery. nPR is defined as having features of CR but with lymphoid nodules in the marrow. PR is defined as ≥50% decrease in ≥2 of the following: lymph nodes, liver and/or spleen size, lymphocytes PLUS ≥1 of the following met: platelets ≥100 x 10^9/L or >50% increase from screening, hemoglobin ≥11 g/dL or >50% increase from screening, CLL cells or B lymphoid nodules in marrow.
ORR per International Workshop on Waldenström's Macroglobulinemia (IWWM) Criteria 2014 as Assessed by the Investigator | Up to ~ 35 months
  ORR per IWWM criteria 2014 is defined as the percentage of participants achieving a CR, very good partial response (VGPR), or PR. CR is defined as all lymph nodes are normal in size (none ≥15 mm), liver and spleen normal in size, serum immunoglobulin M (IgM) values in the normal range, disappearance of monoclonal protein by immunofixation (confirmation needed with a second immunofixation at any subsequent timepoint), and no histological evidence of BM involvement. VGPR is defined as ≥50% decrease from baseline in sum of product of diameter (SPD) of lymph nodes (if abnormal at baseline) ≥50% decrease from baseline in the abnormal portion of the spleen (if previously abnormal) and ≥90% decrease from baseline in serum IgM or serum IgM values in normal range. PR is defined as ≥50% decrease from baseline in SPD of lymph nodes (if abnormal at baseline) ≥50% decrease from baseline in serum IgM and ≥50% decrease from baseline in the abnormal portion of the spleen (if previously abnormal).
ORR per Lugano Criteria 2014 as Assessed by the Investigator | Up to ~ 35 months
  ORR per Lugano criteria 2014 is defined as the percentage of participants achieving a CR or PR. CR defined as EITHER CR by imaging (computed tomography [CT]): all lymph nodes normal (none ≥15 mm) and normal liver and spleen OR complete metabolic response (CMR): assessing fluorodeoxyglucose (FDG) metabolic activity in lymphomatous lesions AND bone marrow normal by morphology. PR defined as EITHER PR by imaging (CT) with ≥50% decrease in the SPD of target lesions, no worsening of nontarget lesions, no new lesions and ≥50% spleen abnormal portion OR Partial Metabolic Response (PMR) with no new lesions and decreased overall uptake AND residual BM abnormalities; OR CR by imaging with residual BM abnormalities; OR PR by imaging without residual BM abnormalities.
Duration of Response (DOR) per iwCLL Criteria 2018 as Assessed by the Investigator | Up to ~ 35 months
  For participants with CR, CRi, nPR, or PR per iwCLL 2018 criteria, DOR is defined as the time from the first documented evidence of objective response until disease progression or death due to any cause, whichever occurs first. CR is defined as meeting the following criteria: no lymph nodes ≥1.5 cm, spleen size <13 cm, liver normal; no constitutional symptoms, normal lymphocyte count, platelets ≥100 x 10^9/L; hemoglobin ≥11 g/dL; and normocellular marrow (no CLL cells or B lymphoid nodules). CRi is defined as meeting CR criteria but with hypocellular bone marrow. nPR is defined as having features of CR but with lymphoid nodules in the marrow. PR is defined as ≥50% decrease in ≥2 of the following: lymph nodes, liver and/or spleen size, lymphocytes PLUS ≥1 of the following met: platelets ≥100 x 10^9/L or >50% increase from screening, hemoglobin ≥11 g/dL or >50% increase from screening, CLL cells or B lymphoid nodules in marrow.
DOR per IWWM Criteria 2014 as Assessed by the Investigator | Up to ~ 35 months
  For participants with CR, VGPR, or PR per IWWM criteria 2014, DOR defined as the time from first documented evidence of objective response until PD or death due to any cause, whichever occurs first. CR defined as all lymph nodes normal in size (none ≥15 mm), liver and spleen normal in size, serum IgM values in normal range, disappearance of monoclonal protein by immunofixation (confirmation needed with second immunofixation at any subsequent timepoint), and no histological evidence of BM involvement. VGPR defined as ≥50% decrease from baseline in SPD of lymph nodes (if abnormal at baseline), ≥50% decrease from baseline in abnormal portion of the spleen (if previously abnormal), and ≥90% decrease from baseline in serum IgM, or serum IgM values in normal range. PR is defined as ≥50% decrease from baseline in SPD of lymph nodes (if abnormal at baseline), ≥50% decrease from baseline in serum IgM, and ≥50% decrease from baseline in abnormal portion of the spleen (if previously abnormal).
DOR per Lugano Criteria 2014 as Assessed by the Investigator | Up to ~ 35 months
  For participants with CR or PR per Lugano criteria 2014, DOR is defined as the time from the first documented evidence of objective response until PD or death due to any cause, whichever occurs first. CR defined as EITHER CR by imaging (CT): all lymph nodes normal (none ≥15 mm) and normal liver and spleen OR CMR: assessing FDG metabolic activity in lymphomatous lesions AND BM normal by morphology. PR defined as EITHER PR by imaging (CT) with ≥50% decrease in the SPD of target lesions, no worsening of nontarget lesions, no new lesions and ≥50% spleen abnormal portion OR PMR with no new lesions and decreased overall uptake AND residual BM abnormalities; OR CR by imaging with residual BM abnormalities; OR PR by imaging without residual BM abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (5):
- China (5):
  - Guangdong Provincial People's Hospital-hematology department ( Site 1002), Guangzhou, Guangdong
  - SUN YAT-SEN UNIVERSITY CANCER CENTRE-Internal medicine ( Site 1007), Guangzhou, Guangdong
  - Henan Cancer Hospital-hematology department ( Site 1003), Zhengzhou, Henan
  - Hunan Cancer Hospital ( Site 1004), Changsha, Hunan
  - Institute of hematology&blood disease hospital-Hematology ( Site 1001), Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/